CLINICAL TRIAL: NCT04834323
Title: Short Term Outcome Of Distal Mesogastric Fixation After Laparoscopic Sleeve Gastrectomy; A Randomized Control Trial
Brief Title: Short Term Outcome Of Distal Mesogastric Fixation After Laparoscopic Sleeve Gastrectomy;
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Said Mohamed Said Abdou Negm, lecturer of general surgery, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Said Negm
Record Dates: First submitted 2021-03-26; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Bariatric Surgery Candidate
Keywords: Laparoscopic Sleeve Gastrectomy

STUDY DESIGN:
Intervention Model Description: This study included patients who were admitted to our center to do laparoscopic sleeve gastrectomy . Cases were collected in the period from December 2019 to December 2020. Sample size was 84 patients divided into 2 equal groups . Group 1: included 42 patients who were subjected to distal mesogastric fixation after laparoscopic sleeve gastrectomy. Group 2: included 42 patients who were subjected to laparoscopic sleeve gastrectomy alone without distal mesogastric fixation.
Masking Description: no masking
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group (1) (Active Comparator): included 42 patients who were subjected to distal mesogastric fixation after laparoscopic sleeve gastrectomy
  Interventions: Procedure: distal mesogastric fixation after sleeve gastrectomy
- group (2) (No Intervention): included 42 patients who were subjected to laparoscopic sleeve gastrectomy alone without distal mesogastric fixation

INTERVENTIONS:
Procedure: distal mesogastric fixation after sleeve gastrectomy — Investigators performed traditional laparoscopic sleeve gastrectomy then we fixed the greater omentum & mesocolon that were cut during gastrectomy to the remaining gstric pouch along the new greater curvature as high as possible along the stable line then we plicated the remaining staple line till angle of His. (the greater omentum & mesocolon not reach this part of staple line) , so the remaining gastric pouch remained tension free and was returned to original position and this may prevent the axial gastric rotation
  Arms: group (1)

SUMMARY:
This study included patients who were admitted to investigator's center to do laparoscopic sleeve gastrectomy . Cases were collected in the period from December 2019 to December 2020. Sample size was 84 patients divided into 2 equal groups . Group 1: included 42 patients who were subjected to distal mesogastric fixation after laparoscopic sleeve gastrectomy. Group 2: included 42 patients who were subjected to laparoscopic sleeve gastrectomy alone without distal mesogastric fixation.

DETAILED DESCRIPTION:
Laparoscopic sleeve gastrectomy is one of weight loss operations and widely performed all over the world . although its widely performed ,it has serious complications like leakage and bleeding . The proposed etiology behind leakage after laparoscopic sleeve gastrectomy may be the axial rotation of the stomach owing to loss of abdominal ligament fixation along the greater curvature of the stomach . The mechanism of increased intra-gastric pressure due to axial gastric rotation may put a lot of stress on the staple lines with increased incidence of leakage. Other complications may occur such as vomiting, food intolerance or persistent reflux.

Objectives:

To assess the effect of distal mesogastric fixation after laparoscopic sleeve gastrectomy to minimize gastric axial rotation and subsequent leakage and other related complications.

Patients and methods:

investigators included all patients who were subjected to laparoscopic sleeve gastrectomy at investigators' center between December 2019 to December 2020. The study was approved by the research and Ethics committee of our university and performed in accordance with the code of ethics of the world medical association (Declaration of Helsinki) for studies involving humans. A written informed consent was obtained from all participants.

Sample size The sample size was calculated using open Epi program using the following data ; confidence interval 95% , power of test 80% , the percent of patients without leak after LSG was 66.6% while after new technique expected to be 95% , odd ratio 9.5% and ratio between two group 1:1; so the calculated sample size was 72 patients , taking into consideration 20% drop outs so the final sample size will be 84 patients divided into 2 equal groups . Group 1: included 42 patients who were subjected to distal mesogastric fixation after laparoscopic sleeve gastrectomy. Group 2: included 42 patients who were subjected to laparoscopic sleeve gastrectomy alone without distal mesogastric fixation.

Patients who had no contraindication for laparoscopic surgery (such as patients with no history of abdominal operations), good general condition with American society of anesthesiology (ASA) I & II, and patients with body mass index above 35 were included. investigators excluded patients who had bad general condition (ASA ≥3), patients with gastro esophageal reflux or hiatal hernia.

Perioperative measures:

In this prospective randomized control trials , all patients were subjected to the followings: patients were selected by randomization method , Full history taking , Complete physical examination , laboratory investigations ( complete blood picture , liver and kidney functions , coagulation profile ) , radiological investigations ( chest x- ray , CT with oral and I.V contrast ) & patients were subjected to upper GI endoscopy.

Surgical techniques :

investigators performed traditional laparoscopic sleeve gastrectomy then investigators fixed the greater omentum & mesocolon that were cut during gastrectomy to the remaining gstric pouch along the new greater curvature as high as possible along the stable line then we plicated the remaining staple line till angle of His. (the greater omentum & mesocolon not reach this part of staple line) , so the remaining gastric pouch remained tension free and was returned to original position and this may prevent the axial gastric rotation as in figures .

Follow up after surgery and discharge from the hospital:

investigators examined the patients clinically, made routine laboratory investigations , made follow up CT with oral and I.V contrast in first week after the operation if suspected leakage & patients were subjected to upper GI endoscopy in first week after the operation if suspected leakage. The patients were followed up for one week, two weeks and one month, 6months post operatively.

Statistical analysis:

The collected data were analyzed by computer using Statistical Package of Social Services version 22 (SPSS), Data were represented in tables and graphs, Continuous Quantitative variables e.g. age were expressed as the mean ± SD & (range), and categorical qualitative variables were expressed as absolute frequencies (number) & relative frequencies (percentage).

Suitable statistical tests of significance were used after checked for normality. Categorical data were cross tabulated and analyzed by the Chi-square test or Fisher's Exact Test; Continuous data were evaluated by student t- test. The results were considered statistically significant when the significant probability was less than 0.05 (P < 0.05). P-value < 0.001 was considered highly statistically significant (HS), and P-value ≥ 0.05 was considered statistically insignificant (NS).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who had no contraindication for laparoscopic surgery.
2. patients with good general condition with American society of anesthesiology (ASA) I & II.
3. patients with body mass index above 35 were included.

Exclusion Criteria:

1 - patients who had bad general condition (ASA ≥3). 2- patients with gastro esophageal reflux or hiatal hernia.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Efficacy of distal mesogasric fixation after laparoscopic sleeve gastrectomy in prevention of Axial gastric rotation. | Within one week after the operation
  Incidence of Axial gastric rotation after the operation
Efficacy of distal mesogasric fixation after laparoscopic sleeve gastrectomy in prevention of gastric leakage . | Within one week after the operation
  Percentage of patients developed gastric leakage after the operation

SECONDARY OUTCOMES:
Quality of life after distal mesogasric fixation after laparoscopic sleeve gastrectomy | Within one month after the operation
  Incidence of side effects of distal mesogasric fixation after laparoscopic sleeve gastrectomy e.g bleeding , vomiting.

CONTACTS AND LOCATIONS:
Overall Officials: Said Mohamed Negm, MD, Principal Investigator — ZAGAZIG UNIVERSITY HOSPITALS
Locations (1):
- Zagazig University Hospitals, Zagazig, Sharqua, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Angrisani L, Santonicola A, Iovino P, Vitiello A, Higa K, Himpens J, Buchwald H, Scopinaro N. IFSO Worldwide Survey 2016: Primary, Endoluminal, and Revisional Procedures. Obes Surg. 2018 Dec;28(12):3783-3794. doi: 10.1007/s11695-018-3450-2. PMID 30121858
- [Background] Benedix F, Poranzke O, Adolf D, Wolff S, Lippert H, Arend J, Manger T, Stroh C; Obesity Surgery Working Group Competence Network Obesity. Staple Line Leak After Primary Sleeve Gastrectomy-Risk Factors and Mid-term Results: Do Patients Still Benefit from the Weight Loss Procedure? Obes Surg. 2017 Jul;27(7):1780-1788. doi: 10.1007/s11695-017-2543-7. PMID 28078641
- [Background] Abou Rached A, Basile M, El Masri H. Gastric leaks post sleeve gastrectomy: review of its prevention and management. World J Gastroenterol. 2014 Oct 14;20(38):13904-10. doi: 10.3748/wjg.v20.i38.13904. PMID 25320526
- [Background] Gagner M. Decreased incidence of leaks after sleeve gastrectomy and improved treatments. Surg Obes Relat Dis. 2014 Jul-Aug;10(4):611-2. doi: 10.1016/j.soard.2014.04.002. Epub 2014 Apr 14. No abstract available. PMID 25224165
- [Background] Nimeri A, Ibrahim M, Maasher A, Al Hadad M. Management Algorithm for Leaks Following Laparoscopic Sleeve Gastrectomy. Obes Surg. 2016 Jan;26(1):21-5. doi: 10.1007/s11695-015-1751-2. PMID 26071239
- [Background] Alizadeh RF, Li S, Inaba C, Penalosa P, Hinojosa MW, Smith BR, Stamos MJ, Nguyen NT. Risk Factors for Gastrointestinal Leak after Bariatric Surgery: MBASQIP Analysis. J Am Coll Surg. 2018 Jul;227(1):135-141. doi: 10.1016/j.jamcollsurg.2018.03.030. Epub 2018 Mar 30. PMID 29605723
- [Background] Parikh M, Issa R, McCrillis A, Saunders JK, Ude-Welcome A, Gagner M. Surgical strategies that may decrease leak after laparoscopic sleeve gastrectomy: a systematic review and meta-analysis of 9991 cases. Ann Surg. 2013 Feb;257(2):231-7. doi: 10.1097/SLA.0b013e31826cc714. PMID 23023201
- [Background] Al-Sabah S, Ladouceur M, Christou N. Anastomotic leaks after bariatric surgery: it is the host response that matters. Surg Obes Relat Dis. 2008 Mar-Apr;4(2):152-7; discussion 157-8. doi: 10.1016/j.soard.2007.12.010. Epub 2008 Mar 4. PMID 18294924
- [Derived] Negm S, Amin M, Shafiq A, Atef B, Yassin M, Farag A. The short-term outcome of distal mesogastric fixation after laparoscopic sleeve gastrectomy: a randomized controlled trial. Surg Today. 2022 Mar;52(3):510-513. doi: 10.1007/s00595-022-02459-x. Epub 2022 Jan 31. PMID 35099602